CLINICAL TRIAL: NCT05509972
Title: International, Prospective, Longterm Study Comparing the Clinical Outcome and In-vivo Wear Behaviour of AS Coated Versus Uncoated Columbus® Total Knee Prosthesis
Brief Title: In-vivo Wear Behaviour of AS Coated Versus Uncoated Columbus® Total Knee Prosthesis
Acronym: COLRAS
Status: Terminated | Type: Observational
Why Stopped: Recruitment too slow
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2024
Record Dates: First submitted 2022-08-11; First posted 2022-08-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Knee Arthritis; Knee Osteoarthritis; Primary Osteoarthritis of Knee Nos; Secondary Osteoarthritis of Knee Nos; Rheumatoid Arthritis of Knee; Instability, Joint; Osteonecrosis; Deformity Knee
Keywords: Total Knee Arthroplasty; Implant Wear; Advanced Surface
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Instability; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Columbus® DD Primary CoCr: Columbus® Deep Dish (DD) Primary Cobalt Chromium (CoCr)
  Interventions: Device: total knee prosthesis implantation
- Columbus® DD Primary CoCr AS coated: Columbus® Deep Dish (DD) Primary Cobalt Chromium (CoCr) Advanced Surface
  Interventions: Device: total knee prosthesis implantation

INTERVENTIONS:
Device: total knee prosthesis implantation — Total Knee Arthroplasty (TKA) represents a well-established, reliable and successful treatment option for end-stage bicompartmental osteoarthritis or comparable conditions even in young patients compromised by knee pain and limitations of daily living
  Other Names: Columbus® Total Knee Arthroplasty

SUMMARY:
This clinical study is a Post-Market Clinical Follow-Up (PMCF) measure and is aiming to compare the in-vivo wear behaviour of the Columbus® total knee prosthesis between the standard Cobalt Chromium (CoCr) and the multilayer coated so called "Advanced Surface" (AS) of the same implant. The clinical investigation is designed as a International, prospective, longterm non-interventional study in order to gain clinical data of many patients within the routine clinical application of the investigational device.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a primary bicondylar total knee endoprosthesis with the Columbus® DD knee prosthesis
* Written signed informed consent of patient
* Willingness and mental ability to participate at the long-term follow-up examinations

Exclusion Criteria:

* Pregnancy
* Patient age <45 and >75years
* Acute inflammatory arthritis
* Coagulation disorders (e.g. Haemophilia)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Polyethylene wear over time | until 10 years postoperatively
  The in-vivo wear of the Polyethylene (PE) tibial tray will be assessed using the observer independent method of the imaging core lab. The PE wear assessment is based on the absolute object position of the knee prosthesis over time.

SECONDARY OUTCOMES:
Implant survival | until 10 years postoperatively
  Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period.
Quality of Life [EQ-5D-5L] compared to baseline | preoperatively and 3 months, 12 months, 2 years, 5 years, 10 years postoperatively
  The 5-dimension 5-level measure of the health status, developed by the EuroQol Group (EQ-5D-5L) is a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
  The answer of each of the five dimensions result in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Progress of Clinical Outcome (Forgotten Joint Score-12) over follow-up period | 3 months, 12 months, 2 years, 5 years, 10 years postoperatively
  The Forgotten Joint Score-12 (FJS-12) Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. These Patient Reported Outcome (PRO) questionnaires focus on patients' awareness of a specific joint in everyday life. In 12 Items the awareness for the artificial joint is assessed by the patient, each on a five point scale (Never / Almost Never / Seldom / Sometimes / Mostly) The Forgotten Joint Score assessment consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Progress of Clinical Outcome [Oxford Knee Score] compared to baseline | preoperatively and 3 months, 12 months, 2 years, 5 years, 10 years postoperatively
  The Oxford Knee Score (OKS) is a reliable 12-item, patient-reported questionnaire originally developed and validated specifically to assess function and pain in patients undergoing total knee replacement. It is short, reproducible, valid and sensitive to clinically important changes over time. Each of the 12 questions on the OKS is scored in the same way with the score decreasing as the reported symptoms increase (i.e. become worse). All questions are laid out with response categories denoting least (or no) symptoms to the left of the page (scoring 4) and those representing greatest severity lying on the right hand side (scoring 0), as detailed for question 1 below. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome,
Radiographic comparison of alignment over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. The radiographic evaluation of Alignment combines Hip-Knee-Angle, femoral and tibial component alignment
Radiographic comparison of implant migration over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. The radiographic evaluation of implant migration comprises tibial and femoral components in m/l and a/p direction,
Radiographic comparison of tibial slope over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. Any changes of Tibial slope over the follow-up period is documented in the radiographic evaluation
Radiographic comparison of the joint line over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine. Any changes of the joint line over the follow-up period is documented in the radiographic evaluation
Adverse events / serious adverse events | During the course of the study up to 10 years postoperatively
  During the course of the study, any upcoming intra- or postoperative (serious) adverse events (AE / SAE) or device effects related or not related to the product under investigation or the procedure, will be documented in the dedicated Case Report Forms. The total number of AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product
Number of Participants with radiological complications over time | During the course of the study up to 10 years postoperatively
  Radiographs shall be standardized between centres as far as possible. Unless limited by patient or equipment constraints, all follow-up imaging examinations will be obtained according to the radiographic protocol of the hospital and the set routine.
  All radiologically evident complications (including fracture, wear, loosening or radiolucencies) are cumulatively documented over the period of follow-up.
Biomechanical analysis of retrievals in case of revision | During the course of the study up to 10 years postoperatively
  Available retrievals of explanted investigational products will be analysed by the biomechanical laboratory of the sponsor according to an analysis protocol which includes the oxidation profile, the wear behaviour, the mechanics and the cumulative linear abrasion of these retrievals.

OTHER OUTCOMES:
Baseline data | preoperatively
  Demographics and medical history
Implant specifications | intraoperatively
  The size and material of each component (tibial and femoral implant, liners, patella resurfacing) of the used implant are documented.
Surgery time | intraoperatively
  the Surgery time from first cut to wound closure is documented
Axis Alignment data according to OrthoPilot® record | intraoperatively
  The orthopaedic navigation system AESCULAP® OrthoPilot® Elite is based on 25 years of experience. During the navigated surgery a record with data on intraoperatively achieved alignment / joint line restoration is stored.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany